CLINICAL TRIAL: NCT03591081
Title: A Feasibility Study to Explore the Implementation and Acceptance of INTELLIN, a Novel mHealth Application on the Management of People With Diabetes Who Have Recently Healed Foot Ulceration.
Brief Title: Induce (Intellin Diabetic Foot) Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natalie Garratt (Other)
Collaborators: Innovate UK (Other Government); Gendius Ltd (Industry)
Responsible Party: Sponsor-Investigator, Natalie Garratt, Research & Development Lead, Northern Care Alliance NHS Foundation Trust
Organization: Northern Care Alliance NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S18DIAB04-S
Record Dates: First submitted 2018-05-31; First posted 2018-07-18 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Healed Ulcer
Keywords: Diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intellin smart phone application (Other): Participants will download a smart phone app, the platform will give the patients daily hints and tips on how to look after their feet.
  Interventions: Other: Intellin smart phone application

INTERVENTIONS:
Other: Intellin smart phone application — This feasibility study will explore if creating an electronic platform Intellin smart phone application can promote and support timely self-referral for individuals with a recently healed DFU. It will explore the software applications acceptance and ease of use for patients.

SUMMARY:
This is a novel feasibility study to test the participant acceptance and usability of a specifically designed smart phone app. It will also explore the effects of smart phone technology in improving self-referrals into the diabetic foot ulcer (DFU) service. Furthermore, it will be explored if this increase in self-referrals will influence the outcome of people with diabetes who have recently had a healed foot ulceration.

DETAILED DESCRIPTION:
The rationale behind this study is if the investigators can introduce a new technology (a smart phone app) which is acceptable to patients, engages them and prompts people to take preventative health behaviours then the investigators may be able to influence the low rates of appropriate self-referral. There is evidence that links poor glycaemic control and hypertension to DFUs, so engagement in these areas of wider diabetes management needs to be reviewed, the latest National Diabetes Audit (NDA) shows only 20% of people with Type 1 and 42% of people with Type 2 diabetes achieve the 3 NICE standards for HbA1c, BP and cholesterol. In addition, healthcare providers are being asked to investigate new systems that may increase patient engagement with and the uptake of the NICE 8 annual care processes. The latest NDA shows only 40% of patients with type 1 and 60% of patients with type 2 diabetes currently have all 8 .

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age will be screened to meet the eligibility criteria:

  * Consultant or GP diagnosis of diabetes mellitus (Type I or II) , documented on the electronic patient record with HbA1C greater than 48mmol/mol
  * History of a recent diabetes foot ulcer defined as being eligible for the national diabetes foot audit and classified as healed for at least 4 weeks and no more than 12 weeks
  * Able to provide informed consent
  * Has no reasons that they could not be part of the study for 12 months such as moving out the area for attending appointments or short life expectancy from a diagnosed illness
  * Owns a smart phone

Exclusion Criteria:

* No smart phone
* Comorbidity such as poor eyesight which limits the use of smart phone
* Participation in an interventional study within the last 30 days
* Critical illness that prevents participating for a period of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
1 Acceptability, suitability and usability of the INTELLIN platform | 12 months
  A 5-point rating scale as assessed by the participants and the clinical team. The 5 point rating is a likert scale where respondants are offered a choice of 5 pre coded responses 1 being strongly disagree 2 disagree 3 (neutral point) niether disagree or agree 4 agree and 5 strongly agree so the individual can express how much they agree or disagree with the experience of using the application
The proportion of patients who self-refer for recurrence of diabetic foot-ulcer over a twelve-month period, compared with the current National diabetes foot audit average of 33.3% | 12 months
  Proportion of participants self-referring using the Intellin platform SOS button over 12 months compared with the current National diabetes foot audit average of 33.3%

SECONDARY OUTCOMES:
Proportion of patients who would recommend Intellin platform to others | 12 months
  A 5-point rating scale as assessed by the participants and the clinical team A 5-point rating scale as assessed by the participants and the clinical team. The 5 point rating is a likert scale where respondants are offered a choice of 5 pre coded responses 1 being strongly disagree 2 disagree 3 (neutral point) niether disagree or agree 4 agree and 5 strongly agree so the individual can express how much they agree or disagree with the experience of using the application.
Proportion of patients who access the Intellin app every day | 12 months
  Case report form and the app electronic database
Proportion of patients who discontinue the study because they are unable to use the app | 12 months
  Case report form
The proportion of patients who report that the INTELLIN app has improved their understanding of the need for the 8 annual checks | 12 months
  Case report form and the app electronic database
The proportion of patients who report that the INTELLIN app has improved their understanding of the management of their diabetes | 12 months
  Case report form and the app electronic database
Proportion of patients completing NICE 8 point annual checks over 12 months compared with the current national diabetes foot audit average of 60% | 12 months
  Case report form and the app electronic database
Proportion of self-referrals that are deemed by the Clinician to be appropriate according to NICE guidelines | 12 months
  Case report form
Time to recurrence of ulcer over 12 months. | 12 months
  Data will be compared to published rates
The impact of using INTELLIN on healthcare utilisation and costs associated with Diabetic Foot Ulcers | 12 months
  Drivers of cost utilisation to include, number of GP visits, outpatient visits, hospital bed medication and type of medication, procedures for patients that develop an ulcer
The effect of using INTELLIN on quality of life | 12 months
  EQ-5D-5L questionnaire
The proportion of patients with recurrence of foot ulcer over 12 months | 12 months
  As compared to published data
The proportion of patients with lower limb amputations | 12 months
  As compared to published data
Changes in cardiovascular markers | 12 months
  Blood pressure measurements, blood test results and medication

CONTACTS AND LOCATIONS:
Overall Officials: Joanne McCardle, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Podiatry Department Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No